CLINICAL TRIAL: NCT03980262
Title: Church, Extension and Academic Partners Empowering Healthy Families
Acronym: EHF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Faith-based partners were not able to recruit sufficient number of families with young children; funding agency approved shift to qualitative study to identify challenges and potential solutions for future faith-partnered health intervention studies.
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Baptist General Convention of Virginia (Unknown); Virginia Cooperative Extension (Unknown); Virginia Family Nutrition Program (Unknown); Virginia Tech Center for Public Health Practice and Research (Unknown)
Responsible Party: Principal Investigator, Kathryn W. Hosig, Associate Professor, Department of Population Health Sciences & Director, Center for Public Health Practice and Research, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017-07071; 2018-68001-27549 (Other Grant/Funding Number: United States Department of Agriculture (NIFA))
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: Obesity; Self-efficacy; Nutrition; Physical Activity; Family-based; Community-Based Participatory Research (CBPR); Faith-based organizations
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Twenty-four churches will participate and each church will be randomly assigned to treatment or control condition. 1) treatment: lifestyle and parenting intervention for parents with a complementary age-appropriate lifestyle curriculum for children and strategies to improve the church health environment (HCHF+); or 2) active control: financial literacy curricula (Money Smart) for parents and children. Churches will receive the alternate program after 12-month data collection for their initial program. This is for community-engaged approach and will also facilitate program evaluation for both the intervention and comparator conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Children, Healthy Families+ (HCHF+) (Experimental): HCHF+ integrates healthful eating and physical activity with parenting education (parent role modeling and child feeding practices) and was recently shown to improve parent and child nutrition behaviors for participants in the Expanded Food and Nutrition Education (EFNEP) program. OrganWise Guys (OWG) will be used for children in first and second grades (ages 6-8). Choose Health: Food, Fun and Fitness (CHFF), developed by Cornell University, will be used for children in grades three through five (ages 8-10). HCHF+ includes 9 sessions to be delivered weekly.
  Interventions: Behavioral: Healthy Children, Healthy Families+ (HCHF+)
- MoneySmart (Active Comparator): A financial education program available through the Federal Deposit Insurance Corporation. Money Smart includes programs for adults and school-aged children, a parent/caregiver guide and a train-the-trainer program. MoneySmart is an Extension-approved program designed to improve money-management practices and financial confidence for parents MoneySmart involves eight weekly sessions that includes one-to-two hour modules with take-home guides for adults. For children, there are eight sessions that include take-home worksheets and a parent/caregiver guide.
  Interventions: Behavioral: Money Smart

INTERVENTIONS:
Behavioral: Healthy Children, Healthy Families+ (HCHF+) — HCHF+ integrates healthful eating and physical activity with parenting education (parent role modeling and child feeding practices) and was recently shown to improve parent and child nutrition behaviors for participants in the Expanded Food and Nutrition Education (EFNEP) program. OrganWise Guys (OWG) will be used for children in first and second grades (ages 6-8). Choose Health: Food, Fun and Fitness (CHFF), developed by Cornell University, will be used for children in grades three through five (ages 8-10). HCHF+ includes 9 sessions to be delivered weekly.
  Arms: Healthy Children, Healthy Families+ (HCHF+)
Behavioral: Money Smart — Money Smart is a financial literacy education program developed by the Federal Deposit Insurance Corporation (FDIC). Curricula are available for both adults and children.
  Arms: MoneySmart

SUMMARY:
The project will address health disparities via a community-engaged approach in partnership with black churches. The long-term goals of this integrated project are to: 1) prevent and reduce childhood obesity through improved parenting practices and home environment related to obesity; 2) expand Extension capacity for community-engaged research and collaborative programming with faith-based organizations; 3) enhance Extension strategies for recruiting and training community volunteers to extend Extension reach; and 4) train future health professionals to provide culturally appropriate collaborative community-based health programs. The project will target the school-aged subset (ages 6-11, first through fifth grade) of the USDA target age range of ages 2-19. The 14-month randomized control trial design of the research component will generate new knowledge regarding effectiveness of a integrated family-based intervention enhanced with social and environmental (church) support to prevent obesity in school-aged children. The research design with a financial literacy active control condition and the primary nutrition and physical activity intervention being tested meets two needs expressed by the community partner and allows rigorous evaluation of both Extension programs. It is hypothesized that parents in the intervention group will have higher levels of self-efficacy for obesity-prevention behaviors, parenting practices related to food and physical activity, improved home food and physical activity. The long term impact is to reduce the prevalence of childhood obesity.

DETAILED DESCRIPTION:
The study follows a group-randomized design. Twenty-four churches will participate based on feasibility and logistical considerations demonstrated in previous work. Church leaders will agree to host the program, identify a church program coordinator to recruit participants and facilitate project implementation, and identify at least two volunteers willing to be trained to deliver the child curricula. Each church will be randomly assigned to treatment condition (HCHF+) or Money-Smart (active control) after baseline data collection. Churches will advertise the Empowering Healthy Families program to church members and to the community at large. The church coordinator will determine the most effective venues and strategies for advertising the program.

Each church will be randomly assigned to one of two treatment conditions: 1) lifestyle and parenting intervention for parents with a complementary age-appropriate lifestyle curriculum for children and strategies to improve the church health environment (HCHF+); or 2) financial literacy curricula (Money Smart) for parents and children (active control). Randomization at the level of church takes advantage of social networking within churches. Consistent with preliminary research, Social Cognitive Theory (SCT), Social-Ecological Model (SEM) and principles of Community based participatory research (CBPR) and community engagement will guide the intervention research and will be reflected in all formative, process and outcome data collection and analyses. Key stakeholders will be involved in all aspects of the research.

Partners include current partners Baptist General Convention of Virginia (BGCVA), Virginia Cooperative Extension's (VCE) Family and Consumer Sciences (FCS) Program at Virginia Tech (VT) and Virginia State University (VSU, historically black state university), Virginia Tech's Center for Public Health Practice and Research (CPHPR) as well as new partners, the Family Nutrition Program (FNP) and 4-H Program at VT and VSU. Partner and Community Involvement in Project Partners and members of the target communities (state, regional and local BGCVA and FNP personnel, church members) will be involved in program planning, implementation, evaluation and sustainability as follows: Identifying strategies to address local strengths, resources, needs and characteristics; Refining strategies to maximize cultural sensitivity for the intervention and research participation, including informed consent documents; Refining strategies to recruit churches/church members and maximize participant retention; Refining program implementation and evaluation plans to maximize program and research fidelity and participation by churches and participants in the education program and data collection; Participating in qualitative data collection during formative and process evaluation; Identifying effective methods to share project outcomes with local and state stakeholders; and Identifying strategies to sustain and expand the program beyond the funding period.

As for data analysis, for qualitative data, a thematic approach will be used to identify themes from semi-structured interviews and focus group discussions. Audio files will be transcribed and transcripts will be reviewed and coded for emergent themes to be checked against field notes. A second researcher will review transcripts, field notes and themes and discrepancies will be rectified. For quantitative data, descriptive univariate analyses will be conducted on all study variables. Data will be checked for outliers, violations of normality and missing data. Predictors of drop-out and non-response will be explored to better understand any discernible systematic processes in play, taking advantage of the data collected until the last time point and demographic variables. If the missingness is found to be random and ignorable, multiple imputations will be used to deal with missing data, else, an intent-to-treat approach that make full use of available data in determining treatment effects will be used for all analyses. Scale scores will be calculated for all outcomes. Because each family (parent-child dyad) is nested within churches, and because there may be more than one parent or more than one child from each family in the program, the investigators will have the advantage of testing family-level effects as well as parent- or child-level effects. A three-level clustered longitudinal model with growth trajectories will be assessed. Quantitative and qualitative outcomes will be triangulated in order to identify the most significant influences on feasibility and sustainability of the interventions and intervention partnerships and on church capacity, readiness, and environment for engaging in health related programming.

ELIGIBILITY:
Inclusion Criteria:

* a parent or primary caregiver and child (age 6-10) dyad living in the same household
* English-speaking

Exclusion Criteria:

* Parent does not have a child between the ages of 6 and 11
* Target child does not live or spend significant time with parent/caregiver
* non-English speaking

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Parental self-efficacy at 6- and 12-months: Self-efficacy for Obesity Prevention Related Behaviors instrument | Baseline, 6-months, 12-months
  Change in parental self-efficacy is measured over time with the 16 item Self-efficacy for Obesity Prevention Related Behaviors Instrument comprised of four validated subscales to assess parent's self-efficacy to help their child get recommended physical activity and fruits and vegetables, and to limit sugary drinks and fruit juice. Specifically, the four subscales are: physical activity (4 items), fruits and vegetables (4 items), sugary drinks (4 items), and fruit juice (4 items). Response options are: not sure, a little sure, sure, very sure, and extremely sure. Scores are summed for each subscale. Scores range from 4 to 20, with higher scores indicating greater self-efficacy (i.e. better outcome).
Change in Child self-efficacy at 6- and 12-months: 3-item response scale | Baseline, 6-months, 12-months
  Change in child self-efficacy is measured over time using procedures validated with 5-10 year old children where pictures of healthy food and physical activity choices are paired with a 3-item response scale: (1) they could not make the healthful choices, (2) they could make the healthful choices sometimes, or (3) they could make the healthful choices all the time. Scores can either be summed or averaged with higher scores indicating greater self-efficacy to make healthful choices (i.e. better outcome).
Change in parental feeding practices/self-regulatory behaviors at 6- and 12-months | Baseline, 6-months, 12-months
  Change in parental feeding practices/self-regulatory behaviors is measured over time using the 31 item Child Feeding Questionnaire uses a 5-point Likert-type scales with responses across seven factor-based domains: perceived responsibility (3 items), perceived parent weight (4 items), perceived child weight (3 items), concern about child weight (3 items), restriction (8 items), pressure to eat (4 items), and monitoring (3 items). Response options vary for each subscale. Means are calculated for each domain. Scores range from 1 to 5 with higher scores indicating higher levels of each domain.
Change in parental supportive behaviors for children's physical activity at 6- and 12-months | Baseline, 6-months, 12-months
  Change in supportive behaviors by parents to enable child physical activity is measured over time with 8 items from the Activity Support Scale (ASS). A 4-point response scale measures parent support for children's physical activity, family co-participation in physical activity, and parent encouragement of child outdoor play. Response options are the following: strongly disagree, disagree, agree, strongly agree.The scale has been shown to be sensitive to change related to a community-based intervention in a similar population as is targeted in the study. The mean is calculated, with possible scores ranging from 1 to 4. Higher scores indicate greater levels of support for physical activity (i.e. better outcome)
Change in home food and physical activity environment at 6- and 12-months | Baseline, 6-months, 12-months
  Change in home food and physical activity environment is measured over time with the Healthy Children, Healthy Families Behavior Checklist (HCHF-BC) developed for use with low-income parents of 3- to 11-year old children. The checklist has demonstrated good reliability (test-retest r=0.83) and convergent validity (scores significantly correlated with validated measures of diet, parent modeling, physical activity and home environment). Six subscales measured are the following: fruits and vegetables, low-fat dairy foods, soda, energy-dense foods, physical activity, and parenting practices. Response options for each item vary. For each individual item, higher values indicate higher frequency of the corresponding behavior. Authors of the instrument recommended computing mean across the items so that higher scores reflect more healthful practices - for this, behaviors or foods that reduced frequency is recommended, the checklist item should be reverse coded in the mean score.

SECONDARY OUTCOMES:
Change in parent nutrition behaviors at 6- and 12-months | Baseline, 6-months, 12-months
  Change in parent nutrition behaviors is measured over time with the validated Block Alive Fat-Sugar-Fruit Vegetable Screener which includes 55 questions and takes about 10-12 minutes. There are two subscales: meat/snacks and fruits/vegetables. For meat and snacks, response options are the following: Once per month or less, 2-3 times per month, 1-2 times per week, 3-4 times per week, and 5 or more times per week. Scores are summed and range from 0 to 60, with higher scores representing greater meat/snack intake. For fruits and vegetables, response options are the following: less than once per week, about once per week, 2-3 times per week, 4-6 times per week, every day, 2 or more times per day. Scores are summed and range from 0 to 35, with higher scores representing greater fruit/vegetable intake.
Change in parent physical activity at 6- and 12-months | Baseline, 6-months, 12-months
  Change in parent physical activity is measured over time with the Godin Leisure-Time Exercise Questionnaire. Weekly frequencies of strenuous, moderate, and mild activities are multiplied by nine, five, and three metabolic equivalents, respectively, and summed to form a measure of total leisure activity. Interpretation of the scoring is the following: 24 unites or more = Active, 14 - 23 = moderately active, Less than 14 unites = insufficiently Active/Sedentary.
Change in child nutrition at 6- and 12-months | Baseline, 6-months, 12-months
  Change in child nutrition is measured over time using the After School Student Questionnaire (ASSQ), which includes questions about child food choices. Constructs measured include: dietary intake for the previous day (6 items), healthy dietary behaviors (6 items), food knowledge (10 items), nutrition knowledge (3 items), food intentions (8 items), and dietary self-efficacy (8 items). Response options vary for each item. For knowledge items, the percentage of correct responses are summed. Higher scores indicated greater knowledge (i.e. better outcome). For behavior and self-efficacy, mean or sum scores are calculated with higher scores indicating higher behavior frequency and high self-efficacy (i.e. better outcome)
Change in child sedentary behavior and physical activity at 6- and 12-months | Baseline, 6-months, 12-months
  Change in child sedentary behavior and physical activity is measured over time using the After School Student Questionnaire (ASSQ), which includes questions about mild and moderate levels of physical activity and physical activity self-regulation. Specific subscales include: physical activity self-efficacy (4 items), participation in sports activities (2 items), and participation in sedentary activities (4 items). For physical activity subscales, sum scores are calculated with higher scores indicating higher frequency of the behavior and self-efficacy (i.e. better outcome). For sedentary behavior, sum scores are calculated with higher scores indicating higher sedentary behavior (i.e. worse outcome)
Change in Child and Parent Body Mass Index (BMI) at 6- and 12-months | Baseline, 6-months, 12-months
  Change in Child and Parent Body Mass Index (BMI) is measured over time without shoes to the nearest ¼ inch using a portable stadiometer. Weight will be measured in light clothing without shoes to the nearest 0.2 pound using a portable digital scale. BMI z-score is recommended for child obesity prevention research. BMI will be calculated from measured height and weight (kg/M2). The better outcome would to see a decrease in BMI for those overweight or obese.

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist General Convention of Virginia, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright JA, Adams WG, Laforge RG, Berry D, Friedman RH. Assessing parental self-efficacy for obesity prevention related behaviors. Int J Behav Nutr Phys Act. 2014 Apr 22;11:53. doi: 10.1186/1479-5868-11-53. PMID 24750693
- [Background] Edmundson E, Parcel GS, Feldman HA, Elder J, Perry CL, Johnson CC, Williston BJ, Stone EJ, Yang M, Lytle L, Webber L. The effects of the Child and Adolescent Trial for Cardiovascular Health upon psychosocial determinants of diet and physical activity behavior. Prev Med. 1996 Jul-Aug;25(4):442-54. doi: 10.1006/pmed.1996.0076. PMID 8812822
- [Background] Edmundson E, Parcel GS, Perry CL, Feldman HA, Smyth M, Johnson CC, Layman A, Bachman K, Perkins T, Smith K, Stone E. The effects of the child and adolescent trial for cardiovascular health intervention on psychosocial determinants of cardiovascular disease risk behavior among third-grade students. Am J Health Promot. 1996 Jan-Feb;10(3):217-25. doi: 10.4278/0890-1171-10.3.217. PMID 10163302
- [Background] Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. Appetite. 2001 Jun;36(3):201-10. doi: 10.1006/appe.2001.0398. PMID 11358344
- [Background] Davison KK, Li K, Baskin ML, Cox T, Affuso O. Measuring parental support for children's physical activity in white and African American parents: the Activity Support Scale for Multiple Groups (ACTS-MG). Prev Med. 2011 Jan;52(1):39-43. doi: 10.1016/j.ypmed.2010.11.008. Epub 2010 Nov 25. PMID 21111755
- [Background] Dickin KL, Hill TF, Dollahite JS. Practice-based evidence of effectiveness in an integrated nutrition and parenting education intervention for low-income parents. J Acad Nutr Diet. 2014 Jun;114(6):945-950. doi: 10.1016/j.jand.2013.09.029. Epub 2013 Dec 4. PMID 24315130
- [Background] Dickin KL, Lent M, Lu AH, Sequeira J, Dollahite JS. Developing a measure of behavior change in a program to help low-income parents prevent unhealthful weight gain in children. J Nutr Educ Behav. 2012 Jan-Feb;44(1):12-21. doi: 10.1016/j.jneb.2011.02.015. Epub 2011 Oct 13. PMID 21996430
- [Background] Block G, Gillespie C, Rosenbaum EH, Jenson C. A rapid food screener to assess fat and fruit and vegetable intake. Am J Prev Med. 2000 May;18(4):284-8. doi: 10.1016/s0749-3797(00)00119-7. PMID 10788730
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Kelder S, Hoelscher DM, Barroso CS, Walker JL, Cribb P, Hu S. The CATCH Kids Club: a pilot after-school study for improving elementary students' nutrition and physical activity. Public Health Nutr. 2005 Apr;8(2):133-40. doi: 10.1079/phn2004678. PMID 15877906
- [Background] Hoelscher DM, Day RS, Kelder SH, Ward JL. Reproducibility and validity of the secondary level School-Based Nutrition Monitoring student questionnaire. J Am Diet Assoc. 2003 Feb;103(2):186-94. doi: 10.1053/jada.2003.50031. PMID 12589324
- [Background] Inokuchi M, Matsuo N, Takayama JI, Hasegawa T. BMI z-score is the optimal measure of annual adiposity change in elementary school children. Ann Hum Biol. 2011 Nov;38(6):747-51. doi: 10.3109/03014460.2011.620625. PMID 22014004
- [Background] Massey OT. A proposed model for the analysis and interpretation of focus groups in evaluation research. Eval Program Plann. 2011 Feb;34(1):21-8. doi: 10.1016/j.evalprogplan.2010.06.003. Epub 2010 Jul 3. PMID 20655593
- [Background] Creswell JW. Qualitative inquiry & research design: Choosing among five approaches (2nd ed). SAGE: Thousand Oaks, CA. 2007
- [Background] Strauss A. Qualitative analysis for social scientists. Cambridge University Press: Cambridge, England. 1987
- [Background] Raykov T. Analysis of longitudinal studies with missing data using covariance structure modeling with full-information maximum likelihood. Structural Equation Modeling.12: 493-505. 2005